CLINICAL TRIAL: NCT02238665
Title: CLE for Differential Diagnosis of IBD
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Helmut Neumann, Professor, University of Erlangen-Nürnberg Medical School
Other Study IDs: HN-0005
Record Dates: First submitted 2014-09-09; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

GROUPS / COHORTS (2):
- Ulcerative colitis
  Interventions: Device: Endomicroscopy
- Crohn's disease
  Interventions: Device: Endomicroscopy

INTERVENTIONS:
Device: Endomicroscopy

SUMMARY:
Differential diagnosis between Ulcerative Colitis (UC) and Crohn's disease (CD) is of pivotal importance for the management of Inflammatory Bowel Disease (IBD) as both entities involve specific therapeutic management strategies. Confocal Laser Endomicroscopy (CLE) allows on demand in vivo characterization of architectural and cellular details during endoscopy. Here, we assessed the efficacy of CLE to differentiate between UC and CD.

ELIGIBILITY:
Inclusion Criteria:

* equal or above 18 years of age
* ability to provide written informed consent
* well-established diagnosis of CD or UC

Exclusion Criteria:

* history of IBD reclassification in the last 3 years
* Boston Bowel Preparation Scale score's < 2 in at least one of the three broad regions of the colon (i.e. rectum plus left side colon, transverse colon plus left and right flexures, right colon)
* inability to provide written informed consent
* severe uncontrolled coagulopathy
* impaired renal function
* pregnancy or breast feeding
* active gastrointestinal bleeding
* known allergy to fluorescein
* residence in institutions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with well-established diagnosis of Crohn's disease and ulcerative colitis.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2009-10; Primary Completion 2013-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with IBD | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Neumann, Professor, Principal Investigator — University Hospital Erlangen
Locations (1):
- University Hospital Erlangen, Erlangen, Germany

REFERENCES:
- [Derived] Tontini GE, Mudter J, Vieth M, Atreya R, Gunther C, Zopf Y, Wildner D, Kiesslich R, Vecchi M, Neurath MF, Neumann H. Confocal laser endomicroscopy for the differential diagnosis of ulcerative colitis and Crohn's disease: a pilot study. Endoscopy. 2015 May;47(5):437-43. doi: 10.1055/s-0034-1391226. Epub 2014 Dec 18. PMID 25521573